CLINICAL TRIAL: NCT03911908
Title: Impact of a NIRS-guided Cardiopulmonary Resuscitation Algorithm Compared to the Current ERC-guideline Algorithm on ROSC Rate and Patient Outcome After In-hospital and Out-of-hospital Cardiac Arrest
Brief Title: Impact of NIRS-guided Cardiopulmonary Resuscitation After Cardiac Arrest on Resuscitation Rate
Acronym: NICA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dr. Serge Thal (Other)
Responsible Party: Sponsor-Investigator, Dr. Serge Thal, Principal Investigator, Johannes Gutenberg University Mainz
Organization: Johannes Gutenberg University Mainz (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-13666; U1111-1231-2797 (Registry Identifier: UTN)
Record Dates: First submitted 2019-04-08; First posted 2019-04-11 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Cardiac Arrest; Cardiopulmonary Arrest With Successful Resuscitation; Cerebral Oxygenation
Keywords: near-infrared spectroscopy; cardiopulmonary resuscitation; cardiac arrest; cerebral oximetry
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: Does near-infrared spectroscopy (NIRS) technology based advanced cardiac life support improve cardiopulmonary resuscitation (CPR) quality in patients (in-house [IHCA] and out-of-hospital cardiac arrest [OHCA], randomized enrollment immediately with CPR) and thereby improve return of spontaneous circulation (ROSC) rate (primary outcome) and patient outcome compared to European Resuscitation Council (ERC)-based CPR (concealed NIRS recording).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: On group will have NIRS reading available to adjust CPR interventions, whereas the control group will not be able use NIRS readings (masked by cover)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ERC guided CPR (intervention/NIRS group) (Active Comparator): CPR protocol according to current ERC guidelines (2015)
  Interventions: Combination Product: Cerebral oximetry (near infrared) based CPR-Algorithm
- ERC-based CPR (control group) (No Intervention): modified CPR protocol based on current ERC guidelines (2015), extended by evaluation of NIRS readings and interventions to optimize CPR quality

INTERVENTIONS:
Combination Product: Cerebral oximetry (near infrared) based CPR-Algorithm — If NIRS values do not increase over time until ROSC (target: >40 % after 10 min), interventions are suggested in a modified CPR/NIRS algorithm.
  Arms: ERC guided CPR (intervention/NIRS group)

SUMMARY:
Sudden cardiac death is one of the main causes of morbidity and mortality worldwide. Cardiac arrest requires prompt intervention by cardiopulmonary resuscitation (CPR). The resuscitation guidelines are the current recommendations for CPR and are revised by expert panels such as the "European Resuscitation Council (ERC)".

Up to now, a parameter for assessing the quality of CPR is missing and further monitoring methods are urgently needed.

Near-infrared spectroscopy (NIRS) is a portable method for measuring regional oxygen levels in the brain. Recent clinical trials suggest that cerebral oxygenation measured by NIRS may correlate with survival and outcome after cardiac arrest.

The investigators propose that NIRS technology may not only be suitable to determine or predict the outcome of the patients, but could also be a useful tool to guide the CPR providers to optimize the CPR techniques and guide the individual treatments/interventions.

The present study was therefore designed to determine if NIRS guided CPR with the aim to optimize NIRS values is superior compared to the current standard practice according to published CPR guidelines (return of spontaneous circulation [ROSC] rate, short and long-term cerebral performance).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a cardiac arrest from the age of 18 years (in and out-of-hospital cardiac arrest)

Exclusion Criteria:

* post-traumatic cardiac arrest
* non-fitting NIRS sensor (size)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-05-22 (Actual); Study Completion 2023-05-05 (Estimated)

PRIMARY OUTCOMES:
successful cardiopulmonary resuscitation (CPR) | DAY 1
  Influence of the intervention on the number of patients with successful return of spontaneous circulation (ROSC) during cardiopulmonary resuscitation (CPR) [ROSC: yes/no]

SECONDARY OUTCOMES:
Time-to-ROSC | DAY 1
  Time from start of cardiopulmonary resuscitation (CPR) until successful return of spontaneous circulation (ROSC) [min]
Cerebral Performance Category (CPC) after successful return of spontaneous circulation (ROSC) | DAY 30, DAY 180, DAY 360
  Neurofunctional recovery, total score, range: 1-5
Glasgow Outcome Scale Extended (GOS-E) after successful return of spontaneous circulation (ROSC) | DAY 30, DAY 180, DAY 360 after successful return of spontaneous circulation (ROSC)
  Neurofunctional recovery, total score, range: 1-8
The Bathel-Index (Barthel) after successful return of spontaneous circulation (ROSC) | Discharge from intensive care unit (variable time point, depending on condition of patient)
  Neurofunctional recovery, total score, range: 0-100

OTHER OUTCOMES:
Neuron Specific Enolase (NSE) blood level after successful return of spontaneous circulation (ROSC) | DAY 1, DAY 2, DAY 3, DAY 4
  NSE as marker for brain damage after cardiac arrest
S100B blood level after successful return of spontaneous circulation (ROSC) | DAY 1, DAY 2, DAY 3, DAY 4
  S100B as marker for brain damage after cardiac arrest
plasminogen activator inhibitor 1/2 (PAI1/2) blood level after successful return of spontaneous circulation (ROSC) after successful return of spontaneous circulation (ROSC) after successful return of spontaneous circulation (ROSC) | DAY 1, DAY 2, DAY 3, DAY 4
  PAI1/2 as marker for brain damage after cardiac arrest
proBNDF/BDNF blood level after successful return of spontaneous circulation (ROSC) | DAY 1, DAY 2, DAY 3, DAY 4
  proBNDF/BDNF as marker for brain damage after cardiac arrest
Neurofilament blood level after successful return of spontaneous circulation (ROSC) | DAY 1, DAY 2, DAY 3, DAY 4
  Neurofilament as marker for brain damage after cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Serge C Thal, MD, Principal Investigator — Department of Anesthesiology
Locations (1):
- Medical Center of the Johannes Gutenberg-University Mainz, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No